CLINICAL TRIAL: NCT00000740
Title: Escalating Multiple-Dose Safety and Tolerance of WR 6026 Hydrochloride in HIV-Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 173; 11148 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; WR 6026
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — 8-aminoquinoline

INTERVENTIONS:
Drug: Sitamaquine

SUMMARY:
To determine the maximum tolerated dose (MTD) of WR 6026 in HIV-infected patients. To determine whether any unexpected toxicities are caused by WR 6026 in HIV-infected patients. To determine whether there is additional toxicity when WR 6026 is given for 21 days rather than 14 days. To further investigate the pharmacokinetics and pharmacodynamics of WR 6026, and in particular to examine potential correlations between the area under the concentration-time curve and methemoglobinemia or other toxicities.

In recent animal studies, WR 6026 demonstrated inhibitory activity against Pneumocystis carinii pneumonia (PCP). This study will assess the safety and tolerance of this drug in HIV-infected patients who do not have PCP.

DETAILED DESCRIPTION:
In recent animal studies, WR 6026 demonstrated inhibitory activity against Pneumocystis carinii pneumonia (PCP). This study will assess the safety and tolerance of this drug in HIV-infected patients who do not have PCP.

Escalating doses of WR 6026 will be studied in successive patient cohorts. Four patients will be randomized to active drug or placebo in a 3:1 ratio at each dose level until moderate toxicity is demonstrated. If one patient at a given dose level experiences WR 6026-related moderate or worse toxicity, the sample size for all subsequent dose levels will be doubled. If two or more patients at a given dose level experience moderate or dose-limiting toxicity, an additional four patients (randomized in the same 3:1 ratio) will be entered at that level, and sample size at all subsequent dose levels will be doubled. Dose escalation will continue until three of six patients receiving active drug at a given dose level experience dose-limiting or worse toxicity, or until two of six patients at a given dose level experience life-threatening toxicity. The MTD will be defined as the dose immediately below the highest dose studied. Eight additional patients will be studied at the presumed MTD to confirm tolerance.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV antibody positive.
* CD4 cell counts less than 500/mm3.
* Adequate general health.
* No significant deterioration in performance status within the past month.
* Prior treatment with a stable regimen of antiretroviral medication for at least 4 weeks prior to study.

Prior Medication:

Required:

* Stable regimen of antiretroviral medication for at least 4 weeks prior to study entry.

Allowed:

* Aerosolized pentamidine for PCP prophylaxis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Intercurrent infection.
* Clinically significant abnormality on EKG.
* Known hypersensitivity to quinolines.
* Known hemoglobin M abnormality.
* Known NADH methemoglobin reductase deficiency.
* Positive test for G6PD deficiency.
* Fever.

Prior Medication:

Excluded:

* Other systemic medication (other than AZT, ddC, ddI, methadone, acyclovir, and NSAIDs) within 3 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Study Completion 1993-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petty BG, Study Chair
Locations (2):
- United States (2):
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland

REFERENCES:
- [Background] Petty BG, Black JR, Hendrix CW, Lewis LD, Basiakos Y, Feinberg J, Pattison DG, Hafner R. Escalating multiple-dose safety and tolerance study of oral WR 6026 in HIV-infected subjects: AIDS clinical trials group 173. J Acquir Immune Defic Syndr. 1999 May 1;21(1):26-32. doi: 10.1097/00126334-199905010-00004. PMID 10235511